CLINICAL TRIAL: NCT01768897
Title: An Open Label, Dose-Escalation Study to Evaluate Safety, Tolerability, Maximum Tolerated Dose (MTD), Efficacy, and Pharmacokinetics (PKs) of CPI-613 Given With High Dose Cytarabine and Mitoxantrone in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: CPI-613, Cytarabine, and Mitoxantrone Hydrochloride in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00022138; NCI-2012-02768 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA012197 (NIH); CCCWFU 22112 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2013-01-11; First posted 2013-01-16 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — devimistat; Cytarabine; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CPI-613, cytarabine, mitoxantrone hydrochloride) (Experimental): Patients receive CPI-613 IV over 2 hours on days 1-5, cytarabine IV over 3 hours every 12 hours for 5 doses beginning on day 3, and mitoxantrone hydrochloride IV over 15 minutes after the 1st, 3rd, and 5th doses of cytarabine. Treatment repeats every 14 days for up to 2 courses* in the absence of disease progression or unacceptable toxicity.
  NOTE: *Patients undergoing a second course of therapy receive CPI-613 IV over 2 hours on days 1-3, cytarabine IV over 3 hours every 12 hours for 5 doses beginning on day 2, and mitoxantrone hydrochloride IV over 15 minutes after the 1st and 3rd doses of cytarabine.
  Interventions: Drug: CPI-613; Drug: cytarabine; Drug: mitoxantrone hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: CPI-613 — Given IV
  Other Names: alpha-lipoic acid analogue CPI-613
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Novantrone
Other: laboratory biomarker analysis — Optional correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of CPI-613 when given together with cytarabine and mitoxantrone hydrochloride in treating patients with relapsed or refractory acute myeloid leukemia. Drugs used in chemotherapy, such as CPI-613, cytarabine and mitoxantrone hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. CPI-613 may help cytarabine and mitoxantrone hydrochloride work better by making cancer cells more sensitive to the drugs

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and maximum tolerated dose (MTD) of CPI-613 when administered with high dose cytarabine, and mitoxantrone (mitoxantrone hydrochloride).

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetics (PKs) of CPI-613 following intravenous (IV) administration in combination with high dose cytarabine and mitoxantrone.

II. To observe the response rate (complete response [CR], complete response with incomplete platelet recovery [CRi] and partial response [PR]) of CPI-613 in combination with high dose cytarabine and mitoxantrone.

III. To observe the overall survival of patients treated with CPI-613 in combination with high dose cytarabine and mitoxantrone.

OUTLINE: This is a dose-escalation study of CPI-613.

Patients receive CPI-613 intravenously (IV) over 2 hours on days 1-5, cytarabine IV over 3 hours every 12 hours for 5 doses beginning on day 3, and mitoxantrone hydrochloride IV over 15 minutes after the 1st, 3rd, and 5th doses of cytarabine. . Treatment repeats every 14 days for up to 2 courses* in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients undergoing a second course of therapy receive CPI-613 IV over 2 hours on days 1-3, cytarabine IV over 3 hours every 12 hours for 5 doses beginning on day 2, and mitoxantrone hydrochloride IV over 15 minutes after the 1st and 3rd doses of cytarabine.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented relapsed and/or refractory acute myeloid leukemia
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 3
* Expected survival > 3 months
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation; (Note: Pregnant patients are excluded because the effects of CPI-613 on a fetus are unknown)
* Fertile men must practice effective contraceptive methods during the study period, unless documentation of infertility exists
* Mentally competent, ability to understand and willingness to sign the informed consent form
* No radiotherapy, treatment with cytotoxic agents (except CPI-613), treatment with biologic agents or any anti-cancer therapy within the 2 weeks prior to treatment with CPI-613; patients must have fully recovered from the acute, non-hematological, non-infectious toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment); patients with persisting, non-hematologic, non-infectious toxicities from prior treatment ≤ grade 2 are eligible, but must be documented as such
* Aspartate aminotransferase ([AST]/serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x upper normal limit (UNL), alanine aminotransferase ([ALT]/serum glutamate pyruvate transaminase [SGPT]) =< 3 x UNL (=< 5 x upper limit of normal [ULN] if liver metastases present)
* Bilirubin =< 1.5 x UNL
* Serum creatinine =< 1.5 mg/dL or 133 μmol/L
* International Normalized Ratio or INR must be < 1.5

Exclusion Criteria:

* Serious medical illness, such as significant cardiac disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, pericardial disease or New York Heart Association class III or IV), or severe debilitating pulmonary disease, that would potentially increase patients' risk for toxicity
* Patients with active central nervous system (CNS) or epidural tumor
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease)
* Pregnant women, or women of child-bearing potential not using reliable means of contraception (because the teratogenic potential of CPI-613 is unknown)
* Lactating females because the potential of excretion of CPI-613 into breast milk (Note: Lactating females are excluded because the effects of CPI-613 on a nursing child are unknown)
* Fertile men unwilling to practice contraceptive methods during the study period
* Life expectancy less than 3 months
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
* Unwilling or unable to follow protocol requirements
* Patients with large and recurrent pleural or peritoneal effusions requiring frequent drainage (e.g. weekly); patients with any amount of clinically significant pericardial effusion
* Active heart disease including myocardial infarction within previous 6 months, symptomatic coronary artery disease, uncontrolled arrhythmias, or symptomatic congestive heart failure
* Albumin < 2.0 g/dL or < 20 g/L
* Evidence of ongoing, uncontrolled infection
* Patients with known human immunodeficiency virus (HIV) infection; (Note: Patients with known HIV infection are excluded because patients with an immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, and because there may be unknown or dangerous drug interactions between CPI-613 and anti-retroviral agents used to treat HIV infections)
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication within the past 2 weeks prior to initiation of CPI-613 treatment (the use of Hydrea is allowed)
* Patients who have received immunotherapy of any type within the past 4 weeks prior to initiation of CPI-613 treatment
* Requirement for immediate palliative treatment of any kind including surgery
* Patients that have received a chemotherapy regimen with stem cell support in the previous 6 months
* A history of additional risk factors for torsade de pointes (e.g., clinically significant heart failure, hypokalemia, family history of long QT syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
MTD of CPI-613 based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE 3.0) | 14 days

SECONDARY OUTCOMES:
Response rate (CR, CRi, and PR) | Day 14 of course 1
  Confidence intervals will be calculated.
Overall survival | Up to 6 months
  We will use Kaplan-Meier estimation.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pardee, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States